CLINICAL TRIAL: NCT05360732
Title: Redefining The Use Of A FOLFIRINOX-Like Regimen In the Front Line In Older Patients With Metastatic Pancreatic Cancer
Brief Title: Redefining FOLFIORINOX in Older Pancreatic Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-1027; GI-170 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2022-04-14; First posted 2022-05-04 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: FOLFIRINOX (Experimental): FOLFIRINOX: Oxaliplatin, Leucovorin and 5-Fluorouracl, Irinotecan,
  Interventions: Drug: FOLFIRINOX

INTERVENTIONS:
Drug: FOLFIRINOX — Alternating FOLFOX and FOLFIRI administered via intravenous infusion. FOLFOX: Oxaliplatin 85 mg/m2 on Day 1; Leucovorin 400 mg/m2 on day 1; 5-FU: 400 mg/m2 IV push on Day 1 followed by 2400 mg/m2 continuous infusion over 46-48 hours. FOLFIRI: Irinotecan 180 mg/m2 on day 1, leucovorin 400 mg/m2, 5-FU: 400 mg/m2 IV push on Day 1 followed by 2400 mg/m2 continuous infusion over 46-48 hours

SUMMARY:
This is a multi- centered two-stage Pilot Study assessing the tolerability and toxicity of an alternating regimen of FOLFOX and FOLFIRI for the treatment of newly diagnosed and untreated metastatic pancreatic cancer in patients over the age of 65 years.

DETAILED DESCRIPTION:
This is a multi-centered two-stage Pilot Study assessing the tolerability and toxicity of an alternating regimen of FOLFOX and FOLFIRI for the treatment of newly diagnosed and untreated metastatic pancreatic cancer in patients over the age of 65 years. Treatment will be given in the outpatient infusion room or clinical research unit. Reported adverse events and potential risks of these agents are described below. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's malignancy.

The study will accrue 37 patients who will be evaluated by correlating their daily activity via use of FitBit that will be provided to the patients, blood markers and progression of the disease with the toxicity grades observed during the treatment. Patients will be treated with standard of care doses of all the chemotherapeutic drugs. The study will be analyzed for futility after treatment of 20 patients. Each cycle consists of 28 days during which patient treatment will alternate between FOLFOX and FOLFIRI on day 1 and day 14 respectively. Patients will be treated until disease progression or any of the conditions listed in Section 4.4 that applies. Patient's response to treatment will be evaluated by CT scans every 8 weeks and the tumor will be assessed using RECIST v1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older
2. The treating physician will use their discretion when assessing if the patient is eligible for this treatment.
3. Patients must have newly diagnosed and previously untreated, histologically or cytologically confirmed adenocarcinoma of the pancreas, with at least one site of metastatic disease (local recurrences after surgery allowed), with lesions that are measurable by RECIST v1.1 criteria. In patients with mixed histology tumors, the predominant feature must be adenocarcinoma.
4. Eastern Cooperative Oncology Group Performance status of 0-2.
5. Previous surgery, adjuvant chemotherapy and/or radiation therapy will be allowed, provided radiation therapy is completed at least 2 weeks prior to signing consent and adjuvant therapy was administered more than 6 months prior to signing consent.
6. Patients must have bone marrow and organ function as defined below:

   * Absolute Neutrophil Count ≥ 1,500/μL
   * Platelets ≥ 100,000/μL
   * Total Bilirubin ≤2 X ULN
   * AST(SGOT)/ALT(SGPT)/

     o Alkaline Phasphatase ≤3 X ULN

     o Or ≤5x ULN if liver metastasis present
   * Creatinine ≤2.0 mg/dL And
   * eGFR (using Cockcroft Gault equation) > 40ml/min
7. Patients must be fluent in English and must be able and willing to undergo Comprehensive Geriatric Assessment
8. Chemotherapy is harmful to the human fetus. For this reason, sexually active males with partners of childbearing potential must agree to use an accepted and effective method of contraception prior to study entry and for the duration of the study.
9. Patients must demonstrate ability to understand and the willingness to sign a written informed consent document.
10. Men and women, regardless of race, ethnic group or sexual orientation are eligible for this study.

Exclusion Criteria:

1. Endocrine or acinar pancreatic carcinoma

2 Patients who have had any systemic chemotherapy in the metastatic or locally advanced inoperable setting (adjuvant or neoadjuvant therapy is allowed)

3 Patients who have received radiation therapy within 2 weeks of signing consent.

4 Patients who are currently receiving or have previously received any other investigational therapy for metastatic pancreatic cancer.

5 Patients with known brain metastases - treated or untreated, are excluded from this study because of their poor prognosis and frequent development of progressive neurological dysfunction that would confound the evaluation of neurologic and other adverse events.

6 Any patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, known HIV-positive patients and those with known active or inactive hepatitis B, untreated HCV or treated HCV without a documented sustained virologic response are excluded from the study.

7 Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active bacterial infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

8 Patients with evidence of active malignancy within 2 years of enrollment without definitive treatment. Patients with localized prostate cancer status-post surgical resection or definitive radiation, localized ER/PR+/HER2- breast cancer status-post definitive local treatment with a low OncotypeDx® on adjuvant hormonal therapy, or local skin cancers that were previously resected will be eligible for inclusion. Patients with a history of in situ cancers treated with definitive local therapy will also be eligible.

9 Patients with grade 3 or higher baseline sensory neuropathy

10 Patients with chronic diarrhea (>4 bowel movements/day) unresolved despite best supportive care for greater than 2 weeks.

11 Patients with any of the following results on the Comprehensive Geriatric Assessment:

* >2 falls in the past month
* BMI <18

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
To assess the toxicity profile of a regimen of alternating FOLFOX and FOLFIRI patients assessed as per NCI's CTCAE v5.0 criteria. | 2 months
  To assess the toxicity profile of a regimen of alternating FOLFOX and FOLFIRI at 2 months in newly diagnosed and untreated metastatic pancreatic adenocarcinoma patients over the age of 65 years deemed ineligible to receive the FOLFIRINOX regimen

SECONDARY OUTCOMES:
To assess the Progression Free Survival (PFS) | 2 years
  To assess the Progression Free Survival (PFS) defined as the time from enrollment to disease progression, death or last patient contact, whichever comes first, for up to 2 years from the end of treatment visit.
To assess the Overall Survival (OS) | 2 years
  Overall Survival (OS) is defined as the time from treatment initiation to death due to any cause or overall survival. Patients will be followed for up to 2 years after the end of treatment visit.
To assess the Objective Response Rate (ORR) | 2 years
  Objective Response Rate (ORR) is defined as the best response in terms of tumor shrinkage measured by RECIST v1.1 criteria obtained during protocol therapy.
To assess the Delayed Toxicity Rate | 8 weeks
  Delayed Toxicity Rate is defined as the absolute percentage of toxicities as measured according toNCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No